CLINICAL TRIAL: NCT00164164
Title: HalfLytely Bowel Prep System for Colonoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: F38-20
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Colonoscopy
Keywords: colonoscopy preparation; prep
MeSH Terms: interventions — polyethylene glycol 3350

INTERVENTIONS:
Drug: HalfLytely
Drug: NuLytely

SUMMARY:
The purpose of the this study was to compare the safety and efficacy of HalfLytely (2L NULYTELY + 20mg bisacodyl) to NULYTELY for preparation prior to colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients at least 18 years of age
* All women of childbearing potential (this includes women who are single and women whose sexual partners have been vasectomized) are required to use medically acceptable contraception during their participation in the study.
* In the investigator's judgment, patient is mentally competent to sign an instrument of informed consent
* Patient is undergoing a colonoscopy for a routinely accepted indication

Exclusion Criteria:

* ileus
* possible intestinal obstruction or perforation
* prior alimentary tract surgery
* significant gastroparesis or gastric outlet obstruction
* impaired consciousness that predisposes a patient to pulmonary aspiration

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 1999-08; Primary Completion 2000-06 (Actual)

PRIMARY OUTCOMES:
Efficacy - Bowel preparation success: preparation rated as "good" or "excellent" by the blinded examiner

SECONDARY OUTCOMES:
Safety - Review of preparation symptoms, adverse events, and laboratory testing

CONTACTS AND LOCATIONS:
Overall Officials: Charles Brady, MD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (2):
- United States (2):
  - Braintree, Massachusetts
  - San Antonio, Texas